CLINICAL TRIAL: NCT04059198
Title: A Phase 2, Exploratory Study Evaluating the Safety and Antiviral Efficacy of Inarigivir Soproxil in Non-cirrhotic Treatment-Naive Subjects Infected With Chronic Hepatitis B Virus
Brief Title: Evaluating the Safety and Efficacy of Inarigivir in Non-cirrhotic Treatment Naive Subjects Infected With Hepatitis B Virus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Evidence of liver injury in a separate Inarigavir study
Sponsor: F-star Therapeutics, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBP-9200-HBV-207
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis B; HBV; Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 - Inarigivir Soproxil Daily (Experimental): Inarigivir Soproxil Alone 400 mg Inarigivir daily for 12 weeks followed by 400 mg daily in combination with TAF 25 mg daily for 12 weeks
  Interventions: Drug: Inarigivir soproxil; Drug: Tenofovir alafenamide fumarate (TAF)
- Arm 2 - Inarigivir Soproxil 3 Times Weekly (Experimental): 400 mg Inarigivir 3 times weekly for 12 weeks followed by 400 mg 3 times weekly in combination with TAF 25 mg daily for 12 weeks
  Interventions: Drug: Inarigivir soproxil; Drug: Tenofovir alafenamide fumarate (TAF)
- Arm 3 - Inarigivir Soproxil and TAF Daily (Experimental): 400 mg Inarigivir daily in combination with TAF 25 mg daily for 24 weeks
  Interventions: Drug: Inarigivir soproxil; Drug: Tenofovir alafenamide fumarate (TAF)

INTERVENTIONS:
Drug: Inarigivir soproxil — Inarigivir soproxil 400 mg tablets
Drug: Tenofovir alafenamide fumarate (TAF) — Tenofovir alafenamide fumarate 25 mg tablet
  Other Names: VEMLIDY

SUMMARY:
An open-label, Phase 2, exploratory study to examine the safety and efficacy of inarigivir in non-cirrhotic, hepatitis B treatment-naive subjects with chronic HBV infection.

ELIGIBILITY:
Inclusion Criteria:

1. HBV-infected male and female subjects aged 18 to 70 years, inclusive
2. Ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI) within 6 months of enrollment date with no evidence of cirrhosis or hepatocellular carcinoma (HCC)
3. Must be willing and able to comply with all study requirements
4. Chronic HBV as defined by documented HBsAg or HBV DNA positive for 6 months or more
5. Not on any antiviral medications for at least 6 months. If a subject is hepatitis B e antigen (HBeAg)-negative, they will be eligible if they have not received antiviral medications for at least 3 months. Antiviral medications include lamivudine, telbivudine, adefovir, tenofovir, entecavir, IFN therapies of any type, and all other medications with potential antiviral activity.
6. HBV DNA >2000 IU/mL for HBeAg-negative subjects and >20,000 IU/mL for HBeAg-positive subjects at Screening
7. ALT <5× ULN and ≤200 U/L
8. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of IP. If the urine pregnancy test is positive, a follow-up serum test is required for confirmation
9. Women of childbearing potential must agree to use a highly effective method of contraception throughout the study and for 3 months after discontinuing study treatment. Men with female partners who are of childbearing potential must agree that they or their partners will use a highly effective method of contraception throughout the study and for 3 months after discontinuing study treatment. Male subjects must not donate sperm throughout the study and for 3 months after discontinuing study treatment.

   * Women of childbearing potential are sexually mature women who have not undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; or who have not been postmenopausal (ie, who have not menstruated at all) for at least 1 year.
   * Highly effective methods of contraception are hormonal contraceptives (oral, injectable, patch, intrauterine devices), male partner sterilization, or total abstinence from heterosexual intercourse, when this is the preferred and usual lifestyle of the subject. Note: The double-barrier method (eg, synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), periodic abstinence (such as calendar, symptothermal, post-ovulation), withdrawal (coitus interruptus), lactational amenorrhea method, and spermicide only are not acceptable as highly effective methods of contraception.
10. Must have the ability to understand and sign a written informed consent form (ICF); consent must be obtained prior to initiation of study procedures

Exclusion Criteria:

1. Any prior liver biopsy evidence of metavir F3 or F4 disease
2. Any history of decompensation of liver disease including history of ascites, encephalopathy, or varices
3. Evidence of advanced fibrosis as defined by Fibroscan at the Screening Visit of ≥8 kPa. If Fibroscan is not available, subjects with both a Fibrotest ≥0.65 and aspartate transaminase (AST):platelet ratio index (APRI) ≥1.0 are excluded (subjects will not be excluded if only 1 of the Fibrotest or APRI results is higher than allowed)
4. Laboratory parameters not within defined thresholds:

   1. White blood cells <4000 cells/μL (<4.0×109/L)
   2. Hemoglobin <11 g/dL (<110 g/L) for females, <13 g/dL (<130 g/L) for males
   3. Platelets <130,000 per μL (<150×109/L)
   4. Albumin <3.5 g/dL (<35 g/L)
   5. International normalized ratio (INR) >1.5
   6. Total bilirubin >1.2 mg/dL (>20.52 μmol/L) or alpha-fetoprotein (AFP) >50 ng/mL (>180.25 nmol/L). Subjects with an elevated indirect bilirubin and known Gilbert's disease can be included if direct bilirubin is within normal limits. Subjects with an AFP >50 ng/mL but <500 ng/mL can be included if CT scan or MRI performed within 3 months shows no evidence of HCC
   7. Creatinine >1.2 mg/dL (>106.08 μmol/L) and creatinine clearance <50 mL/min (<0.83 L/s/m2)
5. Co-infection with hepatitis C virus (HCV), human immunodeficiency virus (HIV), or hepatitis D virus
6. Evidence or history of HCC
7. Malignancy within 5 years prior to Screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible
8. Significant cardiovascular, pulmonary, or neurological disease
9. Received solid organ or bone marrow transplant
10. Received within 3 months of Screening or expected to receive prolonged therapy with immunomodulators (eg, corticosteroids) or biologics (eg, monoclonal antibody, IFN)
11. Subjects currently taking medication(s) that are transported through organic anion transporting polypeptide 1 (OATP1) including, but not limited to, atazanavir, rifampin, cyclosporine, eltrombopag, gemfibrozil, lopinavir/ritonavir, and saquinavir
12. Use of another investigational agent within 3 months of Screening
13. Current alcohol or substance abuse judged by the Investigator to potentially interfere with compliance
14. Females who are pregnant or may wish to become pregnant during the study
15. If the Investigator believes the prospective subject will not be able to comply with the requirements of the protocol and complete the study
16. Any medical condition that, in the opinion of the Investigator, could interfere with evaluation of the study objectives or safety of the subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects reporting an adverse event, clinically significant adverse event, or laboratory abnormality | 24 to 52 weeks
  Proportion of subjects reporting an adverse event or experiencing a clinically significant adverse event or laboratory abnormality from start of treatment to end of inarigivir treatment and 30 days after stopping inarigivir
Percentage of subjects with a ≥1 log10 reduction in HBV DNA, a ≥1 log10 reduction in HBV RNA, and a ≥0.3 log10 reduction in quantitative HBsAg | Baseline to Week 12
  Percentage of subjects with a ≥1 log10 reduction in HBV DNA, a ≥1 log10 reduction in HBV RNA, and a ≥0.3 log10 reduction in quantitative hepatitis B surface antigen (HBsAg) from Baseline to Week 12.
Percentage of subjects with a ≥1 log10 reduction in HBV DNA, a ≥1 log10 reduction in HBV RNA, and a ≥0.5 log10 reduction in quantitative HBsAg | Baseline to Week 24
  Percentage of subjects with a ≥1 log10 reduction in HBV DNA, a ≥1 log10 reduction in HBV RNA, and a ≥0.5 log10 reduction in quantitative hepatitis B surface antigen (HBsAg) from Baseline to Week 24.

SECONDARY OUTCOMES:
Change from Baseline in serum levels of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 | Week 4
  Fold change from Baseline in serum levels of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 at Week 4
Change from Baseline in serum levels of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 | Week 12
  Fold change from Baseline in serum levels of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 at Week 12
Change from Baseline in serum levels of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 | Week 24
  Fold change from Baseline in serum levels of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 at Weeks 24
Change from Baseline in serum levels of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 | Week 48
  Fold change from Baseline in serum levels of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 at Weeks 48
Percentage of subjects who have a ≥0.5 log10 reduction in HBsAg | Week 12
  Percentage of subjects who have a ≥0.5 log10 reduction in hepatitis B surface antigen (HBsAg) at Week 12
Percentage of subjects who have a ≥0.5 log10 reduction in HBsAg | Weeks 24
  Percentage of subjects who have a ≥0.5 log10 reduction in hepatitis B surface antigen (HBsAg) at Week 24
Percentage of subjects with undetectable HBV DNA and HBV RNA | Week 24
  Percentage of subjects with undetectable hepatitis B virus (HBV) DNA and HBV RNA at Week 24
Percentage of subjects with ≥1 log10 reduction in HBsAg | Week 24
  Percentage of subjects with ≥1 log10 reduction in hepatitis B surface antigen (HBsAg) at Week 24
Percentage of subjects with undetectable HBV DNA and HBV RNA | Week 48
  Percentage of subjects with undetectable hepatitis B virus (HBV) DNA and HBV RNA at Week 48
Percentage of subjects with normal ALT | Week 48
  Percentage of subjects with normal alanine aminotransferase (ALT) at Week 48
Percentage of Subjects who were HBeAg-positive at Baseline with loss of HBeAg | Week 24
  Percentage of Subjects who were hepatitis B e-antigen (HBeAg)-positive at Baseline with loss of HBeAg at Week 24
Percentage of Subjects who were HBeAg-positive at Baseline with loss of HBeAg | Week 48
  Percentage of Subjects who were hepatitis B e-antigen (HBeAg)-positive at Baseline with loss of HBeAg at Week 48
Percentage of Subjects who were HBeAg-positive at Baseline with > 0.5 log10 reduction in HBeAg | Week 12
  Percentage of Subjects who were hepatitis B e-antigen (HBeAg)-positive at Baseline with > 0.5 log10 reduction in HBeAg at Week 12
Percentage of Subjects who were HBeAg-positive at Baseline with > 0.5 log10 reduction in HBeAg | Week 24
  Percentage of Subjects who were hepatitis B e-antigen (HBeAg)-positive at Baseline with > 0.5 log10 reduction in HBeAg at Week 24
Percentage of Subjects who were HBeAg-positive at Baseline with > 0.5 log10 reduction in HBeAg | Week 48
  Percentage of Subjects who were hepatitis B e-antigen (HBeAg)-positive at Baseline with > 0.5 log10 reduction in HBeAg at Week 48
Percentage of Subjects who were HBeAg-positive at Baseline with > 1 log10 reduction in HBeAg | Week 12
  Percentage of Subjects who were hepatitis B e-antigen (HBeAg)-positive at Baseline with > 1 log10 reduction in HBeAg at Week 12
Percentage of Subjects who were HBeAg-positive at Baseline with > 1 log10 reduction in HBeAg | Week 24
  Percentage of Subjects who were hepatitis B e-antigen (HBeAg)-positive at Baseline with > 1 log10 reduction in HBeAg at Week 24
Percentage of Subjects who were HBeAg-positive at Baseline with > 1 log10 reduction in HBeAg | Week 48
  Percentage of Subjects who were hepatitis B e-antigen (HBeAg)-positive at Baseline with > 1 log10 reduction in HBeAg at Week 48
Percentage of Subjects who enter the Long-term Follow-up Period with undetectable HBV DNA and HBV RNA | Week 72
  Percentage of Subjects who enter the Long-term Follow-up Period with undetectable heaptitis B virus (HBV) DNA and HBV RNA at Week 72
Percentage of Subjects who enter the Long-term Follow-up Period who remain HBV DNA <2000 IU | Week 72
  Percentage of Subjects who enter the Long-term Follow-up Period who remain hepatitis B virus (HBV) DNA <2000 IU at Week 72
Percentage of Subjects who enter the Long-term Follow-up Period with HBsAg loss | Week 72
  Percentage of Subjects who enter the Long-term Follow-up Period with hepatitis B surface antigen (HBsAg) loss at Week 72
Percentage of Subjects who enter the Long-term Follow-up Period with normal ALT | Week 72
  Percentage of Subjects who enter the Long-term Follow-up Period with normal alanine aminotransferase (ALT) at Week 72
Percentage of Subjects who enter the Long-term Follow-up Period who were HBeAg-positive at Baseline with loss of HBeAg | Week 72
  Percentage of Subjects who enter the Long-term Follow-up Period who were hepatitis B e-antigen (HBeAg)-positive at Baseline with loss of HBeAg at Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Don Mitchell, Study Director — Spring Bank Pharmaceuticals
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong, Hong Kong Island
  - Prince of Wales Hospital, Shatin, New Territories